CLINICAL TRIAL: NCT06687252
Title: Ancillary Study of Retrospective Analysis of Neonatal Management of Patients with ANtenatal Diagnosis of Variation of Genital Development At Lyon Hospital
Brief Title: Retrospective Analysis of the Neonatal Management of Patients with an Antenatal Diagnosis of Genital Development Variation At the Hospital of Lyon
Acronym: PECAN-VDG
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_5313
Record Dates: First submitted 2024-05-21; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-05

CONDITIONS: Endocrinology; Disorders of Sexual Development; Prenatal Diagnosis; Psychology; Gonadal Dysgenesis; Androgen Abnormalities; Hypospadias; Bladder Extrophy; Androgen Overproduction; Gonadal Development Abnormalities; Turner Syndrome; Klinefelter's Syndrome; Mixed Gonadal Dysgenesis; Ovotestis; Chimera
Keywords: Endocrinology; Disorders of Sexual Development; Prenatal diagnosis; Psychology; Gonadal dysgenesis; Androgens; Hypospadias; Bladder extrophy; Sexual development; Turner syndrome; Klinefelter's syndrome; Gonadal dysgenesis, mixed; Ovotesticular disorders of sex development; Chimera
MeSH Terms: conditions — Disorders of Sex Development; Gonadal Dysgenesis; Hypospadias; Bladder Exstrophy; Turner Syndrome; Klinefelter Syndrome; Gonadal Dysgenesis, Mixed; Ovotesticular Disorders of Sex Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All fetuses referred to the HFME and Croix Rousse CPDPNs for antenatal diagnostic consultation (DAN): Non-interventional retrospective study, only on datas for suspected isolated variation in genital development (VDG)

SUMMARY:
Variations in genital development (VDG) account for 0.5% to 1% of births. Advances in ultrasound techniques, as well as in prenatal diagnosis techniques, particularly in genetics, have led to improvements in the prenatal diagnosis of these pathologies. However, to date, there is no consensus on etiological research and standardized management of these patients and their families, once VDG has been detected.

The value of multidisciplinary management has already been demonstrated, but a number of grey areas remain: the frequency of false-positive ultrasound findings, the place of invasive antenatal diagnostic tests, the role left to parents during the diagnostic process, the frequency of associated malformations discovered post-natally, and how to prepare for immediate management at birth.

The aim of this study is to improve the management of patients and their families as soon as a Disorders of Sexual Development is detected antenatally.

The primary objective is to describe the management, particularly complementary investigations performed in the antenatal management of ultrasound diagnoses of Disorders of Sexual Development over the last 10 years.

The secondary objectives are :

* To determine the correlation between pre- and post-natal morphological phenotype and the proportion of false positives in antenatal ultrasound diagnosis.
* To characterize prenatally diagnosed Disorders of Sexual Development
* To determine the proportion of isolated prenatally-diagnosed Disorders of Sexual Development that turn out not to be isolated during postnatal follow-up.
* The evaluation of the care pathway :

  * To establish the frequency of prenatal psychological support for parents
  * To establish the role of parents in prenatal diagnosis strategy decisions at our center

ELIGIBILITY:
Inclusion Criteria:

Fetuse of the hospital Femme-Mère-Enfant, the hospital Croix Rousse and Lyon-Sud hospital, reffered to Pluridisciplinary Centers for Prenatal Diagnosis (CPDPNs) for antenatal diagnosis (DAN) for a suspected isolated Disorders of Sexual Development (DSD) from January 2013 to December 2022.

Intrauterine growth retardation (RCIU), a muscular or minor ventricular septal defect, or a pyloric dilatation are not considered as an associated malformation.

Exclusion Criteria:

* No follow-up file at the CPDPN of the hospital Femme-Mère-Enfant, the hospital Croix Rousse or of Lyon-Sud hospital.
* Lack of data and identification of the child born.
* Referred to CPDPN for urinary malformation including no VDG.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All fetuses referred to the hospital Femme-Mère-Enfant and the hospital Croix Rousse Pluridisciplinary Centers for Prenatal Diagnosis (CPDPNs), for antenatal diagnosis (DAN) for a suspected isolated Disorders of Sexual Development (DSD) from 01/01/2013 to 31/12/2023.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Ancillary Study of Retrospective Analysis of Neonatal Management of Patients with ANtenatal Diagnosis of Variation of Genital Development at Lyon Hospital | From January 2013 to December 2022.
  Number and type of complementary investigations performed as part of antenatal management following ultrasound diagnoses of Disorders of Sexual Development over the past 10 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'endocrinologie pédiatrique HFME, Bron, France